CLINICAL TRIAL: NCT05992129
Title: Structural Foot Types and Their Influence on Core Strength and Athletic Performance in Collegiate Athletes
Brief Title: Influence of Foot Types on Collegiate Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Magdalena (Other)
Responsible Party: Principal Investigator, Orlando Santiago Moreno Barriga, physician, Universidad del Magdalena
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTUM212170
Record Dates: First submitted 2023-07-14; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: low foot; high foot; performance; core

STUDY DESIGN:
Intervention Model Description: After initial measurements of dependent variables (electromyographic activity amplitude of core muscles, static stability, dynamic stability, ergospirometry, countermovement jump, and 40m sprint test), athletes are divided into two groups: 1) Case group, which is further classified into (a) athletes with high arched feet and (b) athletes with flat feet, and 2) Control group, consisting of athletes with neutral feet. The case group performs intrinsic and extrinsic foot muscle strengthening exercises for 12 weeks, while the control group does not engage in these exercises. Following intervention, both case and control groups are re-evaluated in dependent variables to conduct pre-post intervention variable comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- structural foot types and their influence on core in collegiate athletes (Other): Athletes do 12 weeks of exercises and then evaluate how they influenced core stability
  Interventions: Other: foot exercise
- structural foot types and their influence on performance in collgiate athletes (Other): Athletes do 12 weeks of exercises and then evaluate how they influenced on sport performance
  Interventions: Other: foot exercise

INTERVENTIONS:
Other: foot exercise — These are foot and ankle muscle strengthening exercises described and evaluated by the literature

SUMMARY:
The purpose of the study is to assess whether high or low arch foot types influence the overall performance of the athlete.

DETAILED DESCRIPTION:
After meeting the eligibility criteria for the study, university athletes have their general athletic condition variables evaluated in the laboratory and in the field. Subsequently, athletes with high and low arches perform 12-week foot muscle strengthening exercises to re-evaluate the variables in both athletes with high and low arch types who performed the strengthening exercises, as well as those with neutral arch who did not perform the exercises.

ELIGIBILITY:
Inclusion Criteria:

* University athletes with 4 years of continuous training
* high foot
* low foot.
* Neutral foot

Exclusion Criteria:

* Any pain
* active injuries
* biomechanical alteration in their lower extremities.
* Spine disorders
* Spine surgery
* abdominal surgery,
* neural or vestibular disease
* arthritis of the lower extremities
* used of alcohol, sedatives, pain relievers, cold medication, or stimulants in the last year
* rigid pronated foot

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to the finding that over 80% of university athletes were male and, furthermore, over 70% of those with high or low arches were male, it was decided to conduct the study on men in order to have a significant sample for the study
Enrollment: 97 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Alterations change from baseline of the muscles of the center of gravity at 12 weeks | Baseline and week 12
  Measurement of the activity of the muscles of the center of gravity with electromyography
  1. Voltage amplitude of the anterior rectus muscle measured in millivolts
  2. Erector spinae muscle voltage amplitude measured in millivolts
  3. Voltage amplitude of the external oblique muscle measured in millivolts
  4. Voltage amplitude of the Internal oblique muscle measured in millivolts
  Electrodes were placed on the subjects according to literature recommendations (Oliva-Lozano & Muyor, 2020). Three sets of three exercise repetitions were performed (García-Vaquero et al., 2012).
Alterations change from baseline of static stability: total mean distance, Anterioposterior distance and mediolateral distance at 12 weeks | Baseline and week 12
  The static stability in terms of total mean distance, Anterioposterior distance and mediolateral distance were measured in millimeters.
  The stability was measured when the athlete stood on the dominant leg trying to maintain balance for 10 seconds.
Alterations change from baseline of static stability: total mean speed, anterio-posterior speed and mediolateral speed at 12 weeks | Baseline and week 12
  The static stability in terms of static stability: total mean speed, anterio-posterior speed and mediolateral speed were measured in millimeters/seconds The stability was measured when the athlete stood on the dominant leg trying to maintain balance for 10 seconds.
Alterations change from baseline of static stability: covered area at 12 weeks | Baseline and week 12
  The static stability in terms of static covered area was measured in millimeters² The stability was measured when the athlete stood on the dominant leg trying to maintain balance for 10 seconds.
Alterations change from baseline of dynamic stability: mean power at 12 weeks | Baseline and week 12
  The dynamic stability in terms of mean power was measured in watts/kilogram
  The participants were instructed to perform five single-leg jumps using their dominant foot.
Alterations change from baseline of dynamic stability: left-right and forward/backward displacement at 12 weeks | Baseline and week 12
  The dynamic stability in terms of left-right and forward/backward displacement were measured in centimeters The participants were instructed to perform five single-leg jumps using their dominant foot.
Alterations change from baseline of dynamic stability: covered area at 12 weeks | Baseline and week 12
  The dynamic stability in terms of covered area measured in centimeters² The participants were instructed to perform five single-leg jumps using their dominant foot.
Alterations change from baseline in sport performance of maximum oxygen consumption (VO2max) and anaerobic threshold (AT) at 12 weeks | Baseline and week 12
  We used an Ergospirometry system to assess:
  VO2max and AT measured in milliliters/kilogram/minute
  They followed Marcos' protocol for a continuous treadmill exercise test (Marcos et al., 2018) and estimated VO2max and AT.
Alterations change from baseline in sport performance of countermovement jump test: maximum force measured at 12 weeks | Baseline and week 12
  Sport performance of countermovement jump test: maximum force measured in Newton/kilogram.
  For the countermovement jump (CMJ), participants started upright, knees and hips flexed, and then jumped while crossing their hands behind their back (Bobbert et al., 1996).
Alterations change from baseline in sport performance of countermovement jump test: rate of force development at 12 weeks | Baseline and week 12
  Sport performance of countermovement jump test: rate of force development measured in Newton/kilogram/second.
  For the countermovement jump (CMJ), participants started upright, knees and hips flexed, and then jumped while crossing their hands behind their back (Bobbert et al., 1996).
Alterations change from baseline in sport performance of countermovement jump test: maximum power at 12 weeks | Baseline and week 12
  Sport performance of countermovement jump test: maximum power measured in Watts/kilogram.
  For the countermovement jump (CMJ), participants started upright, knees and hips flexed, and then jumped while crossing their hands behind their back (Bobbert et al., 1996).
Alterations change from baseline in sport performance of countermovement jump test:maximum velocity at 12 weeks | Baseline and week 12
  Sport performance of countermovement jump test: maximum velocity measured in meters/second.
  For the countermovement jump (CMJ), participants started upright, knees and hips flexed, and then jumped while crossing their hands behind their back (Bobbert et al., 1996).
Alterations change from baseline in sport performance of record time 40-meter sprint test at 12 weeks | Baseline and week 12
  Sport performance of of 40-meter sprint test: record time measured in seconds. To measure the 40-meter sprint, photocell sensors and biomechanical equipment were used and participants ran at their maximum speed over a distance of 40 meters
Alterations change from baseline in sport performance of speed 40-meter sprint test at 12 weeks | Baseline and week 12
  Sport performance of of 40-meter sprint test: speed measured in meters/second. To measure the 40-meter sprint, photocell sensors and biomechanical equipment were used and participants ran at their maximum speed over a distance of 40 meters
Alterations change from baseline in sport performance of acceleration 40-meter sprint test at 12 weeks | Baseline and week 12
  Sport performance of of 40-meter sprint test: acceleration measured in meters/second².
  To measure the 40-meter sprint, photocell sensors and biomechanical equipment were used and participants ran at their maximum speed over a distance of 40 meters

CONTACTS AND LOCATIONS:
Overall Officials: orlando santiago Moreno barriga, Principal Investigator — Universidad del Magdalena
Locations (1):
- Universidad del Magdalena, Santa Marta, Magdalena Department, Colombia

REFERENCES:
- [Background] Oliva-Lozano JM, Muyor JM. Core Muscle Activity During Physical Fitness Exercises: A Systematic Review. Int J Environ Res Public Health. 2020 Jun 16;17(12):4306. doi: 10.3390/ijerph17124306. PMID 32560185
- [Background] Garcia-Vaquero MP, Moreside JM, Brontons-Gil E, Peco-Gonzalez N, Vera-Garcia FJ. Trunk muscle activation during stabilization exercises with single and double leg support. J Electromyogr Kinesiol. 2012 Jun;22(3):398-406. doi: 10.1016/j.jelekin.2012.02.017. Epub 2012 Mar 20. PMID 22436839
- [Background] Marcos MA, Koulla PM, Anthos ZI. Preseason Maximal Aerobic Power in Professional Soccer Players Among Different Divisions. J Strength Cond Res. 2018 Feb;32(2):356-363. doi: 10.1519/JSC.0000000000001810. PMID 29369953
- [Background] Bobbert MF, Gerritsen KG, Litjens MC, Van Soest AJ. Why is countermovement jump height greater than squat jump height? Med Sci Sports Exerc. 1996 Nov;28(11):1402-12. doi: 10.1097/00005768-199611000-00009. PMID 8933491

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT05992129/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT05992129/ICF_001.pdf